CLINICAL TRIAL: NCT07275658
Title: Timing and Dose of Fluid Deresuscitation in Critically Ill Patients: a Prospective Observational Multicenter Study
Brief Title: Timing and Dose of Fluid Deresuscitation in Critically Ill Patients
Acronym: TIDE
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: OLVG (Network)
Responsible Party: Principal Investigator, P.R. Tuinman, Prof. Dr. P.R. Tuinman, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2025.0391
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Fluid Overload; Critical Care, Intensive Care; Deresuscitation
Keywords: ultrasound, RRT, furosemide
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fluid deresuscitation is an important intervention in the Intensive Care Unit (ICU). This study aims to find (1) determinants of successful deresuscitation, (2) the optimal rate (dose) of deresuscitation based on these determinants, and (3) differences in metabolic profiles for a more personalized approach of deresuscitation.

This study is a multicenter, prospective, observational cohort study in critically ill patients. This study will include ICU patients who have a clinical indication for deresuscitation as set by the treating physician. Clinical, ultrasound and laboratory values will be collected and used for analysis.

DETAILED DESCRIPTION:
Primary objective:

The aim of this study is to identify determinants of successful deresuscitation in ICU patients, defined as achieving a negative fluid balance within 24 hours without hemodynamic consequences.

Secondary objectives:

* Timing of deresuscitation:

  * Identify determinants of successful deresuscitation in ICU patients, defined as achieving a negative fluid balance within 24 hours;
  * Compare these determinants with determinants for the clinical decision of deresuscitation by the treating physician;
  * Identify differences in these determinants within subgroups of sepsis, ARDS and cardiac patients, provided the numbers are sufficient;
* Rate (dose) of deresuscitation:

  * Identify parameters associated with diuretic or natriuretic response during deresuscitation;
  * Find individualized optimal rates of deresuscitation based on these determinants;
* Possible complications of deresuscitation:

  * Determine whether there is an association between electrolyte or acid-base disturbances during deresuscitation (e.g. the Strong Ion Difference) and clinical outcomes;
  * Determine whether there is an association between the rate of deresuscitation and hemodynamic consequences;
  * Determine whether there is an association between the timing and rate of deresuscitation and atrial fibrillation (AF);
  * Determine whether there is an association between deresuscitation and the occurrence of delirium;
  * Determine whether there is an association between timing and rate of deresuscitation and acute kidney injury (AKI).

Study design:

The TIDE study is a multicenter, prospective, observational cohort study in the ICUs of the Amsterdam UMC and OLVG in Amsterdam, the Netherlands.

Study population:

Adult patients admitted to the ICU, who have a clinical indication for deresuscitation as set by the treating physician, using diuretics or ultrafiltration; first deresuscitation attempt during the ICU stay.

Sample size calculation:

For finding associations with logistic regression with a moderate (odds ratio >1.5) to strong (odds ratio >2.5) effect an alpha set at 0.05, power set at 0.8 and an estimated failure of 50% or more, we would need a sample size of around 150-210 patients.

Methods:

Patients in the participating ICUs are screened for eligibility when the treating physician sets a clinical indication for deresuscitation. Eligible patients will be included in the study. At that time, defined as baseline, clinical, ultrasound and laboratory measures will be collected. Clinical measures among others include: heart rate, mean arterial pressure, dose of vasopressors, and capillary refill time. Ultrasound measurements include: lung ultrasound scores (LUS), venous excess ultrasound (VExUS), and cardiac ultrasound, including VTI during a passive leg raise (PLR). Laboratory measurements include arterial blood gas analysis and urinalysis. Furthermore, baseline characteristics such as demographics, reason for ICU admission, severity of illness scores, and medical history are collected.

Deresuscitation will be performed according to standard care according to the treating physician's insights. Primary follow up is 24 hours in which granular data of deresuscitation tactics, deresuscitation output, electrolyte and acid-base disturbances, and hemodynamic consequences are collected. Secondary follow up is at 7 days for complications such as acute kidney injury and at 28 days for mortality, ICU length of stay (LOS) and ventilator free days (VFD), where available.

ELIGIBILITY:
Inclusion Criteria:

* Admission to one of the participating ICUs;
* Clinical indication for deresuscitation using diuretics or ultrafiltration as set by the treating physician; first attempt during the ICU stay.

Exclusion Criteria:

* Age below 18 years old;
* Major cardiac shunts;
* Moderate to severe aortic regurgitation;
* Morbid Obesisty (BMI >40);
* POCUS impossible or unreliable (i.e. pre-existing interstitial lung disease);
* PLR or modified form of PLR impossible (i.e. ECMO);
* Transfer from another ICU;
* Previous inclusion in this study;
* Patients who are moribund or facing the end of life;
* Opt out.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Successful deresuscitation without hemodynamic consequences | 24 hours
  Reach negative fluid balance in first 24 hours without hemodynamic consequences (yes/no), defined as either hypotension or hypoperfusion:
  1. Hypotension
     * Interventions required to maintain blood pressure MAP > 65mmHg
     * Deresuscitation is stopped
     * Fluid bolus needs to be given
     * Noradrenaline (or other vasopressor) needs to be initiated, increased to > 0.2 microg/kg/min, or increased by 50%
     * Dose reduction or interruption of RRT
  2. Hypoperfusion (one of the following):
     * Arterial lactate level >3 and/or increased 25% or more
     * New development of mottled skin
     * Capillary refill time > 3 seconds
     * New oliguria (urine output < 0.3-0.5ml/kg/hour for the previous 6 hours)

SECONDARY OUTCOMES:
Successful deresuscitation | 24 hours
  Reach negative fluid balance in the first 24 hours
Rate of deresuscitation | 24 hours
  Urine output or ultrafiltration rate in mL/kg/h
Dose of deresuscitation | 24 hours
  Fluid balance in mL/kg
Natriuresis | 24 hours
  Urinary sodium output in mmol/L/24h
Delta Strong Ion Difference | 24 hours
  ΔSID in mmol/L
Delta serum sodium | 24 hours
  Serum ΔNa in mmol/L
Delta serum chloride | 24 hours
  Serum ΔCl in mmol/L
Atrial fibrillation | 24 hours
  Occurrence of ≥1 hour AF or AF for which treatment is needed during the deresuscitation window if not present at baseline
Acute Kidney Injury (AKI) | 7 days
  AKI as diagnosed based on the Kidney Disease Improving Global Outcomes (KDIGO) criteria:
  Stage 1: sCreat 1.5-1.9 times baseline OR ≥0.3 mg/dl (≥26.5 mmol/l) increase OR urine output <0.5 ml/kg/h for 6-12 hours Stage 2: sCreat 2.0-2.9 times baseline OR urine output <0.5 ml/kg/h for ≥12 hours Stage 3: sCreat 3.0 times baseline OR Increase in serum creatinine to ≥4.0 mg/dl (X353.6 mmol/l) OR Initiation of renal replacement therapy OR urine output <0.3 ml/kg/h for ≥24 hours OR anuria for ≥ 12 hours
Persistent AKI | 7 days
  Prolonged AKI for ≥48 hours if not present before start deresuscitation
Renal Replacement Therapy (RRT) | 7 days
  Need for RRT after start deresuscitation if not used at baseline and primary deresuscitation
Delirium | 7 days
  Need 1 or more types of medication to treat delirium after start deresuscitation
ICU-mortality | 28 days
  Mortality within ICU stay
28-day mortality | 28 days
  Mortality after 28 days
Ventilator free days (VFD) | 28 days
  Patient is alive and breathes without assistance of the mechanical ventilator, if the period of unassisted breathing lasted at least 24 consecutive hours:
  * VFD-28 = 0 if subject dies within 28 days of mechanical ventilation
  * VFD-28 = 28 - x if successfully liberated from ventilation x days after initiation successful liberation: extubation (planned or unplanned) without death or reintubation within the next 72 hours
  * VFD-28 = 0 if the subject is mechanically ventilated for ≥ 28 days
ICU length of stay (LOS) | 28 days
  Length of stay in the intensive care unit

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - OLVG, Amsterdam
  - Amsterdam UMC, Amsterdam